CLINICAL TRIAL: NCT00543322
Title: PET Study of the Nicotinic Receptors in Human : Brain Distribution and Quantification
Brief Title: PET Study of the Nicotinic Receptors in Human
Status: Terminated | Type: Observational
Sponsor: Commissariat A L'energie Atomique (Other Government)
Other Study IDs: SHFJ-100008
Record Dates: First submitted 2007-10-11; First posted 2007-10-12 (Estimated); Last update posted 2007-10-12 (Estimated); Status verified 2007-10

CONDITIONS: Healthy; Parkinson Disease; Alzheimer Disease; Epilepsy
MeSH Terms: conditions — Parkinson Disease; Alzheimer Disease; Epilepsy

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to quantify the brain distribution of the nicotinic receptors in human volunteers and their alterations in patients suffering from neurological diseases such as Parkinson and Alzheimer diseases and familial epilepsy. This will be done using Postron Emission Tomography (PET) and a new radiotracer of the nicotinic receptors.

DETAILED DESCRIPTION:
PET is a non -invasive technique that allow to study, in vivo in human, the neurotransmission system. Thanks to the development of radiotracers that are selective for the binding site of the neurotransmitter, several system have been studied such as the dopaminergic, GABAergic system.

However, the in vivo study of the cholinergic system, was hampered the lack of suitable radiotracer. The cholinergic system is an important neurotransmitter system in human brain which exact rule remains unclear. It is involved in cognition, and memory and it is altered early in several neurodegeneratives diseases such as Parkinson and Alzheimer diseases.

The nicotinic receptors are one target of the cholinergic neurotransmission (together with muscarinic receptors), that are of importance since postmortem studies have showed their early alteration in neurodegeneratives diseases. Moreover, as they are located mostly on presynaptic part of the cholinergic terminations, their labelling can be of great interest for the study of the integrity of the cholinergic fibres.

Post-mortem studies have shown a reduction of the nicotinic receptors density in Alzheimer's disease in temporal cortex and hippocampus. Similarly, in Parkinson's diseases, nicotinic receptor density have been shown to be reduced in fronto-temporal cortex and in pedoculo-pontin nuclei. Recently, point mutation on nicotinic receptor sub-units (alpha4 or beta2) have been objectived in a familial epilepsy: the Autosomic Dominant Noctural Frontal Lobe Epilepsy (ADNFLE). Nicotinic receptor are also involved in tobacco addiction, as they are the main brain target of the nicotine from the cigarette smoking. Human post-mortem studies and animal models suggest that nicotinic receptor density is increased in chronic smoker.

The in vivo study of these receptors will bring new insight in the understanding of the physiopathology of nicotinic receptor in several neurodegeneratives diseases.

The radioligand that will be used is the2- F-A-85380 labelled with fluorin-18, a fluoro derivative of the A85380 (Abbott compound). The 2-F-A-85380 present a high affinity and high selectivity for the alpha4beta2 nicotinic receptor subtype, which is the major nicotinic receptor subtype in the brain. Radiolabelling, with fluorin-18 (half-life=110 min) performed in our laboratory, allow produciton of a high specific activity.

This compound has been studied extensively in rodent and in monkey using PET. The low toxicity of this compound allow its use as a radiotracer in human.

Subject between 18 and 85 years of age may be eligible for this study. Candidates are screened with a medical history and physical examination, psychological assessment, and blood and urine tests.

Subjects enrolled in the study participate in one of the following procedures:

Part 1 : Quantification in normal non-smoker and smokers subjects:

Two catheters (small plastic tubes) are placed into veins in the subject's arms for injecting [18F]FA85380 and for collecting blood samples during the scan. A third catheter is placed into a wrist artery to obtain arterial blood during the scan. With the catheters in place, the subject lies down on the scanner bed with his or her head placed in a special mask that limits movement during the brain scan. The scan begins with an initial transmission scan to measure tissue attenuation for about 15 minutes, after which the [18F]FA85380 is injected and the actual PET scan starts. The entire procedure takes about 4 hours, including 2.5 hours of continuous scanning sessions, during which the subject is required to lie still. The second scan period start after one hour rest period where subjects can relax out of the scanner, and last 30 minutes. They are monitored throughout the procedure. Vital signs are measured and electrocardiogram is taken before and after injection of the tracer. At the end of the scanning, additional blood and urine samples are collected. Subjects are asked to urinate after each scanning session to lessen the radioactivity in the body.

Part 2 Parkinson disease :

The PET scan using [18F]FA85380 is the same as in Part 1. A second PET procedure using [18F]FDOPA is performed the day after.

Part 3 Alzheimer disease This part of the study is the same as Part 1, except that no arterial catheter is placed. A second PET procedure is performed using [18F]FDG.

Part 4 Epilepsy ADNFLE This part of the study is the same as Part 3.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion criteria:

* Subjects under 60 years are only male.
* Subjects from 60 to 85 may be male or female
* Subjects that have a Health insurance
* Subjects will be asked to refrain from caffein for at least 12 hours

Specific inclusion criteria for part 2:

* Subjects with

Specific inclusion criteria for part 3:

* Subjects with Alzheimer diseased based on the DSM IV and NINCDS-ADRDA criteria. With a MMS between 15 and 26 (included).
* Subjects capable of giving an informed consent and accompagined by a person of confidence

Specific inclusion criteria for part 4:

* Subjects with ADNFLE with or without demonstrated mutation on the nicotinic receptors

Exclusion Criteria:

General exclusion criteria:

* Subjects with abnormal MRI findings at visual inspection
* Subjects with a history of significant medical disordres, or requiering chronic treatment that interfere with the cholinergic system
* Subjects with abnormal plasma biological analysis
* Subjects with significant past and present history of hypertension, cardiovascular disease and diabetes mellitus
* Subjects who have pacemakers, aneurysm clips (metal clips) metallic prostheses (including heart valves and cochlear implants) or shrapnel fragments.
* Subjects incapable of giving an informed consent

Specific exclusion criteria for part 2:

* Subjects with a smoking history in the last five years

Specific exclusion criteria for part 3:

* Subjects with a smoking history in the last five years

Specific exclusion criteria for part 4:

* Subjects with a smoking history in the last five years

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2001-07; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MICHEL BOTTLAENDER, MD PhD, Principal Investigator — CEA
Locations (1):
- CEA, Service Hospitalier Frederic Joliot, Orsay, France